CLINICAL TRIAL: NCT02859168
Title: Randomized, Single-blind, Placebo-controlled Cross-over Design of Myofascial Induction and Placebo Electrotherapy in Breast Cancer Survivors
Brief Title: Myofascial Induction in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Manuel Arroyo Morales, PhD, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FIS PI10/02749-02764
Record Dates: First submitted 2016-08-01; First posted 2016-08-08 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Pain; Breast Cancer
Keywords: Neck; Shoulder; Manual Therapies
MeSH Terms: conditions — Pain; Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Myofascial Induction session (Experimental): Patients received a Myofascial Induction focused on the upper limb area for 30 minutes using the Pilat approach.
  Interventions: Behavioral: Myofascial Induction
- Placebo session (Placebo Comparator): Patients received a placebo session consisted of 30 minutes of unplugged pulsed shortwave therapy.
  Interventions: Device: Unplugged pulsed shortwave therapy

INTERVENTIONS:
Behavioral: Myofascial Induction — Patients received a Myofascial Induction focused on the upper limb area for 30 minutes using the Pilat approach.
  Arms: Myofascial Induction session
Device: Unplugged pulsed shortwave therapy — Patients received a placebo session consisted of 30 minutes of unplugged pulsed shortwave therapy.
  Arms: Placebo session

SUMMARY:
The purpose of this study was to show the immediate effects of myofascial induction on perceived pain and anxiety, cervical/shoulder range of motion and mood state in breast cancer survivors suffering shoulder/arm morbidity.

DETAILED DESCRIPTION:
Background: To investigate the immediate effects of myofascial induction on perceived pain and anxiety, cervical/shoulder range of motion and mood state in breast cancer survivors suffering shoulder/arm morbidity.

Methods: Randomized, single-blind, placebo-controlled cross-over study. Twenty-one enrolled participants who had a diagnosis of breast cancer stage I-IIIA and had completed adjuvant therapy except hormonal treatment. The study consisted of two intervention sessions of 30 minutes separated by a wash-up period of 4 weeks. The interventions consisted of a Myofascial Induction (experimental group) or placebo pulsed shortwave therapy (control group). The main outcome measures were: Visual Analogue Scale for pain and anxiety, shoulder-cervical goniometry for range of motion, Profile of Mood States for psychological distress and Attitudes Toward Massage Scale.

ELIGIBILITY:
Inclusion Criteria:

* had a diagnosis of breast cancer (cancer stage I-IIIA)
* was between the ages of 25 and 65
* had completed adjuvant therapy except hormonal treatment

Exclusion Criteria:

* had cancer recurrence

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS). Change scores | A wash-up period of 4 weeks between the 2 sessions was established
  A numerical rating scale that contains scores in the range of 0 to 10 (0 = 'no pain/anxiety'; 10 = 'worst imaginable pain/anxiety level'). Participants must mark the level of pain that they feel at that moment in the cervical-arm area and use the scale to indicate their anxiety level.

SECONDARY OUTCOMES:
Goniometry shoulder. Change scores | A wash-up period of 4 weeks between the 2 sessions was established
  A plastic universal goniometer with two adjustable overlapping arms to measure the active range of motion of the shoulder joint.
Goniometry cervical. Change scores | A wash-up period of 4 weeks between the 2 sessions was established
  A cervical goniometric device manufactured by Performance Attainment Associates (St Paul, MN, USA) to measure the active range of motion of the cervical joints.
Profile of Mood States (POMS). Change scores | A wash-up period of 4 weeks between the 2 sessions was established
  This questionnaire is a measure of psychological distress. This questionnaire contains 65 items assessing mood state, which are grouped into six subscales: tension-anxiety, depression-dejection, anger-hostility, vigour-activity, fatigue-inertia and confusion-bewilderment.
Attitudes toward massage (ATOM) scale | Covariates
  The Attitudes toward massage (ATOM) scale is a nine-item measure of overall attitude toward massage composed of the 'Massage as Healthful' and the 'Massage as Pleasant' subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Arroyo-Morales, PhD, Principal Investigator — Deparment of Physical Therapy, Faculty of Health Sciences, University of Granada
Locations (1):
- Faculty of Health Sciences. University of Granada, Granada, Spain

REFERENCES:
- [Result] Castro-Martin E, Ortiz-Comino L, Gallart-Aragon T, Esteban-Moreno B, Arroyo-Morales M, Galiano-Castillo N. Myofascial Induction Effects on Neck-Shoulder Pain in Breast Cancer Survivors: Randomized, Single-Blind, Placebo-Controlled Crossover Design. Arch Phys Med Rehabil. 2017 May;98(5):832-840. doi: 10.1016/j.apmr.2016.11.019. Epub 2016 Dec 18. PMID 28003133